CLINICAL TRIAL: NCT06365034
Title: A Single-center, Retrospective Study on the Efficacy and Safety of Conversion Therapy for Patients With Initially Unresectable Hepatocellular Carcinoma
Brief Title: Study on the Efficacy and Safety of Conversion Therapy in Patients With Initially Unresectable Hepatocellular Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: YKLL-KY-2024（024）
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tumor tissue and adjacent tissues of the patient
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the efficacy and safety of conversion therapy in patients with initially unresectable hepatocellular carcinoma (uHCC).

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of conversion therapy in patients with initially unresectable hepatocellular carcinoma (uHCC). Exon sequencing, 16SrRNA sequencing and immunohistochemistry were used to verify the protein expression, revealing the mechanism of tumor occurrence and development from the genome level, and providing reference for immunotherapy, targeted drug use and curative effect evaluation of tumors.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old, gender is not limited;
* Patients with radiographically or pathologically confirmed, unresectable advanced hepatocellular carcinoma;
* At least one measurable lesion according to the mRECIST criteria as the target lesion;
* No prior immunotherapy, including but not limited to anti-CTLA-4, anti-PD-1, and anti-PD-L1 antibodies;
* Patients with an ECOG score of 0-2 were included according to the activity status score scale developed by the Eastern Cooperative Oncology Group (ECOG) in the United States;
* Child-Pugh liver function is graded as A or B.

Exclusion Criteria:

* Have a history of immunodeficiency, or have other acquired or congenital immunodeficiency diseases;
* Have other malignancies;
* Presence of any active autoimmune disease or history of autoimmune disease (including, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism), or known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation, or other patients who are considered by the investigator to have an impact on study treatment;
* Long-term heavy use of corticosteroids or other immunomodulators;
* Serious illness in combination with other systems;
* Received a live or attenuated vaccine within 30 days prior to the first dose, or plans to receive a live or attenuated vaccine during the study, excluding the new crown vaccine;
* Known human immunodeficiency virus (HIV) infection;
* Have participated in other therapeutic clinical studies;
* Incomplete clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with initial unresectable hepatocellular carcinoma who have undergone conversion therapy.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic response rate | 2 years
  Proportion of patients whose tumors have shrunk to a prespecified value and are able to maintain the minimum time limit

CONTACTS AND LOCATIONS:
Overall Officials: Jing Liang, Dr, Study Director — the Qianfoshan Hospital
Locations (1):
- the Qianfoshan Hospital, Jinan, Shandong, China